CLINICAL TRIAL: NCT06097156
Title: Feasibility Evaluation of See.d Pre-Analytical Platform Performance: From Whole Blood to Plasma and SBS Slides for Liquid Biopsy Applications
Brief Title: Evaluation of See.d as an Automated Blood Sample Preparator for Multiple Liquid Biopsy Applications
Status: Recruiting | Type: Observational
Sponsor: Tethis S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: TET-22-001
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants; Breast Cancer
Keywords: Breast Cancer; Metastatic Patients; Liquid Biopsy; Whole Blood; Plasma; White Blood Cells; Pre-Analytical Standardization
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy donors: Participants who are in good health and without history of cancer disease
- Metastatic Breast Cancer patients: Metastatic breast cancer category is based on the definition of the European Society of Medical Oncology and is defined as disease spread to other parts of the body, such as bones, liver or lungs (also called stage IV). Tumours at distant sites are called metastases.

SUMMARY:
This study aims to evaluate the feasibility of using See.d instrument and SBS slides for preparation of plasma and cytological samples from whole blood.

Forty-five participants will be enrolled (20 healthy volunteers and 25 metastatic breast cancer patients) and each participant will be asked to provide a blood sample.

DETAILED DESCRIPTION:
The goal of this study is the evaluation of a new instrument called See.d, to be used in conjunction with its accessories, Smart Bio Surface (SBS) slides, for preparation of cytological samples (seeded on SBS slides) and plasma from fresh whole blood (within 4-6 hours from collection).

Blood samples collected from healthy volunteers will be spiked-in with reference DNA and mock-CTC to mimic a patient sample in order to evaluate the instrument performance through the analysis of several parameters.

Blood samples from Metastatic Breast Cancer (MBC) patients will be processed with See.d instrument installed in a clinical context to perform a preliminary analytical characterization of either cell-free DNA (cfDNA) and Circulating Tumor Cells (CTC).

For its feasibility nature, no formal statistics has been planned for this study.

ELIGIBILITY:
Inclusion Criteria:

* General (all participants)

  * Participants is willing and able to give and sign a written informed consent
  * Aged 18 or above
* Specific for metastatic breast cancer patients

  * Female for metastatic breast cancer patients, aged 18 or above
  * Histological confirmation of breast cancer
  * Presence of at least one non-bone metastasis
  * Disease assessed to be in clinical or radiologic progression to the last line of treatment, as evaluated by the investigator
  * The biopsy, when recommended by the oncologist, is scheduled within 4 weeks after the date of blood withdrawal
  * Last biopsy or any other minor surgical procedure was perfomed at least 7 days before blood withdrawal
  * Known Bilirubin level ≥ 2 mg/dL on a blood sample collected within 7 days from the enrolment. If unavailable, it is not necessary to assess bilirubin
* Specific for healthy participants

  * Both sexes for healthy volunteers, aged 18 or above
  * Healthy participants who visit the site for reason other than cancer diagnosis (including breast cancer).

Exclusion Criteria:

* Ongoing infections requiring antibiotic or antiviral treatment
* Previous history of a blood cancer or an invasive non-BC apart from cancers treated with curative intent at least 3 years previously with no recurrence since diagnosis with the exception of non-melanoma skin cancer. For healthy participants also includes breast cancer
* Undergone major surgery < 4 weeks prior to the time of blood collection
* Initiated a new line of treatment after disease progression at the time of blood or tissue biopsy collection
* Presence of known severe coagulation or haematological disorder
* Pregnancy
* For metastatic breast cancer patients: histological confirmation of a Triple Negative Breast Cancer (TNBC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from among the people who visit the Breast department
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of White Blood Cells adhered on SBS slides | 1 day (at the blood draw)
  Evaluation of total adhered cell count on SBS slides
SBS slides stability | 1 day (at the blood draw)]
  Evaluation of the area of adhered cell nuclei on SBS slides
cfDNA quality control | 1 day (at the blood draw)
  Evaluation of the ratio between cfDNA and genomic contaminant DNA
Feasibility of using See.d SBS slides for subsequent analysis | 1 day (at the blood draw)
  Recovery of putative Circulating Tumor Cells (CTCs)
Feasibility of using See.d plasma for subsequent analysis | 1 day (at the blood draw)
  Detection of already known DNA mutations

CONTACTS AND LOCATIONS:
Overall Officials: Luca Mazzarella, MD, Principal Investigator — IEO Hospital
Locations (1):
- IEO, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
This is a preliminary research study without an IPD information sharing plan

REFERENCES:
- [Background] Gennari A, Andre F, Barrios CH, Cortes J, de Azambuja E, DeMichele A, Dent R, Fenlon D, Gligorov J, Hurvitz SA, Im SA, Krug D, Kunz WG, Loi S, Penault-Llorca F, Ricke J, Robson M, Rugo HS, Saura C, Schmid P, Singer CF, Spanic T, Tolaney SM, Turner NC, Curigliano G, Loibl S, Paluch-Shimon S, Harbeck N; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. ESMO Clinical Practice Guideline for the diagnosis, staging and treatment of patients with metastatic breast cancer. Ann Oncol. 2021 Dec;32(12):1475-1495. doi: 10.1016/j.annonc.2021.09.019. Epub 2021 Oct 19. No abstract available. PMID 34678411
- [Background] Turashvili G, Brogi E. Tumor Heterogeneity in Breast Cancer. Front Med (Lausanne). 2017 Dec 8;4:227. doi: 10.3389/fmed.2017.00227. eCollection 2017. PMID 29276709
- [Background] Seale KN, Tkaczuk KHR. Circulating Biomarkers in Breast Cancer. Clin Breast Cancer. 2022 Apr;22(3):e319-e331. doi: 10.1016/j.clbc.2021.09.006. Epub 2021 Sep 22. PMID 34756687
- [Background] Ignatiadis M, Sledge GW, Jeffrey SS. Liquid biopsy enters the clinic - implementation issues and future challenges. Nat Rev Clin Oncol. 2021 May;18(5):297-312. doi: 10.1038/s41571-020-00457-x. Epub 2021 Jan 20. PMID 33473219
- [Background] Carbone R, Marangi I, Zanardi A, Giorgetti L, Chierici E, Berlanda G, Podesta A, Fiorentini F, Bongiorno G, Piseri P, Pelicci PG, Milani P. Biocompatibility of cluster-assembled nanostructured TiO2 with primary and cancer cells. Biomaterials. 2006 Jun;27(17):3221-9. doi: 10.1016/j.biomaterials.2006.01.056. Epub 2006 Feb 28. PMID 16504283
- [Background] Krol I, Schwab FD, Carbone R, Ritter M, Picocci S, De Marni ML, Stepien G, Franchi GM, Zanardi A, Rissoglio MD, Covelli A, Guidi G, Scarinci D, Castro-Giner F, Mazzarella L, Doglioni C, Borghi F, Milani P, Kurzeder C, Weber WP, Aceto N. Detection of clustered circulating tumour cells in early breast cancer. Br J Cancer. 2021 Jul;125(1):23-27. doi: 10.1038/s41416-021-01327-8. Epub 2021 Mar 24. PMID 33762721